CLINICAL TRIAL: NCT01936909
Title: Interleukin-1 Blockade in Recently Decompensated Heart Failure: A Randomized Placebo-controlled Double-blinded Study
Brief Title: Interleukin-1 Blockade in Recently Decompensated Heart Failure
Acronym: RED-HART
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RED-HART (HM15339); 1R34HL117026 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Anakinra (short) (Experimental): Anakinra 100 mg daily for 2 weeks, followed by placebo for 10 weeks
  Interventions: Drug: Anakinra (weeks 1-2)
- Anakinra (long) (Experimental): Anakinra 100 mg daily for 12 weeks
  Interventions: Drug: Anakinra (weeks 1-2); Drug: Anakinra (weeks 3-12)
- Placebo (Placebo Comparator): Placebo injections daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra (weeks 1-2) — Anakinra 100 mg daily for weeks 1 and 2
  Arms: Anakinra (long); Anakinra (short)
Drug: Anakinra (weeks 3-12)
  Other Names: Anakinra 100 mg daily for weeks 3 through 12
  Arms: Anakinra (long)
Drug: Placebo
  Other Names: Placebo daily for week 1 through 12
  Arms: Placebo

SUMMARY:
The RED-HART is a randomized double-blinded placebo-controlled study of Anakinra (IL-1 blocker) in patients with recently decompensated heart failure to determine the safety and efficacy in terms of aerobic exercise capacity and ventilatory efficiency measured with a cardiopulmonary exercise test.

ELIGIBILITY:
Inclusion Criteria:

All 6 criteria need to be met for enrollment of the patient in the study

1. Primary diagnosis for hospitalization is decompensated heart failure established as the finding at admission of all 2 conditions listed below:

   1. dyspnea or respiratory distress or tachypnea at rest or with minimal exertion;
   2. evidence of elevated cardiac filling pressure or pulmonary congestion (at least one of the conditions must be met);

      * pulmonary congestion/edema at physical exam OR chest X-Ray;
      * plasma Brain Natriuretic Peptide (BNP) levels ≥200 pg/ml;
      * invasive measurement of left ventricular end-diastolic pressure >18 mmHg or of pulmonary artery occluding pressure (wedge) >16 mmHg.
2. The patient has a prior documentation of impaired left ventricular systolic function (ejection fraction <50%) at most recent assessment by any imaging modality (within 12 months).
3. The patient is now clinically stable and meets standard criteria for hospital discharge as documented by all the 3 conditions listed below:

   1. absence of dyspnea or pulmonary congestion/distress at rest;
   2. absence of pitting edema in the lower extremities, or in any other region;
   3. stable hemodynamic parameters (blood pressure, heart rate).
4. The patient is of age ≥21 years old, and is willing and able to provide written informed consent.
5. The patient is willing and able to comply with the protocol (i.e. self administration of the treatment, and exercise protocol).
6. The patient has screening plasma C-reactive protein levels >2 mg/L.

Exclusion Criteria Subjects will not be eligible if they meet any of the following 15 exclusion criteria.

1. The primary diagnosis for admission is NOT decompensated heart failure, including diagnosis of acute coronary syndromes, hypertensive urgency/emergency, tachy- or brady-arrhythmias.
2. Concomitant clinically significant comorbidities that would interfere with the execution or interpretation of the study including but not limited to acute coronary syndromes, uncontrolled hypertension or orthostatic hypotension, tachy- or brady-arrhythmias, acute or chronic pulmonary disease or neuromuscular disorders affecting respiration.
3. Recent (previous 3 months) or planned cardiac resynchronization therapy (CRT), coronary artery revascularization procedures, or heart valve surgeries.
4. Previous or planned implantation of left ventricular assist devices or heart-transplant.
5. Chronic use of intravenous inotropes.
6. Recent (<14 days) use of immunosuppressive or anti-inflammatory drugs (not including Non-Steroidal Anti-Inflammatory Drugs [NSAIDs]).
7. Chronic inflammatory disorder (including but not limited to rheumatoid arthritis, systemic lupus erythematosus).
8. Active infection (of any type);
9. Chronic/recurrent infectious disease (including Hepatitis B virus [HBV], Hepatitis C virus [HCV], and HIV/AIDS).
10. Prior (within the past 10 years) or current malignancy.
11. Any comorbidity limiting survival or ability to complete the study.
12. End stage kidney disease requiring renal replacement therapy.
13. Neutropenia (<2,000/mm3) or Thrombocytopenia (<50,000/mm3).
14. Pregnancy.
15. Angina, arrhythmias, or electrocardiograph (ECG) changes that limit maximum exertion during cardiopulmonary exercise testing obtained during the baseline testing.

Ages: 21 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University; Benjamin W Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Van Tassell BW, Canada J, Carbone S, Trankle C, Buckley L, Oddi Erdle C, Abouzaki NA, Dixon D, Kadariya D, Christopher S, Schatz A, Regan J, Viscusi M, Del Buono M, Melchior R, Mankad P, Lu J, Sculthorpe R, Biondi-Zoccai G, Lesnefsky E, Arena R, Abbate A. Interleukin-1 Blockade in Recently Decompensated Systolic Heart Failure: Results From REDHART (Recently Decompensated Heart Failure Anakinra Response Trial). Circ Heart Fail. 2017 Nov;10(11):e004373. doi: 10.1161/CIRCHEARTFAILURE.117.004373. PMID 29141858

RESULTS

PARTICIPANT FLOW:
Groups:
- Anakinra (Long): Anakinra 100 mg daily for 12 weeks
  Anakinra (weeks 1-2): Anakinra 100 mg daily for weeks 1 and 2
  Anakinra (weeks 3-12)
- Placebo: Placebo injections daily for 12 weeks
  Placebo
Period: Overall Study
Arm/Group | Anakinra (Short) | Anakinra (Long) | Placebo
Started | 20 | 20 | 20
Completed | 10 | 12 | 14
Not Completed | 10 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra (Short) | Anakinra (Long) | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 15 | 48
  >=65 years | 4 | 3 | 5 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [49.75 to 60.5] | 53.5 [47.25 to 60.75] | 59.5 [56.25 to 66.5] | 56.5 [50.25 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 17
  Male | 15 | 14 | 14 | 43
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Interval Changes in Peak Oxygen Consumption (VO2)
Description: Interval changes in peak oxygen consumption (VO2) after 2 weeks of anakinra treatment.
Time Frame: Baseline to 2 weeks
Population: Patients who completed baseline and 2 week exercise evaluation
Measure: Median (Inter-Quartile Range); unit: mL/kg/min
Arm/Group | Anakinra (Short) | Anakinra (Long) | Placebo
Number analyzed (Participants) | 16 | 18 | 18
mL/kg/min
  Baseline | 14.05 [11.225 to 16.15] | 14.45 [11.075 to 16.575] | 13.3 [11.975 to 15.30]
  2 weeks | 14.85 [12.525 to 16.375] | 14.45 [11.075 to 17.725] | 12.65 [11.575 to 17.025]
Statistical Analysis 1: Comparison: Anakinra (Short) vs Anakinra (Long) vs Placebo; This test reflects a comparison between baseline and 2 weeks (both rows); Test type: Superiority; p > 0.20, ANOVA

2. Secondary Outcome: Quality of Life Improvement
Description: The Duke Activity Status Index questionnaire will be completed at enrollment and 12 weeks. The scale ranges from 0 (unable to perform any tasks) to 58.20 (able to perform all tasks). Higher scores represent increased ability to perform daily activities and may be interpreted as improved quality of life.
Time Frame: 12 weeks
Population: Patients with baseline and follow-up data
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Anakinra (Short) | Anakinra (Long) | Placebo
Number analyzed (Participants) | 16 | 18 | 18
units on a scale
  Baseline | 26.95 [17.325 to 47.2] | 23.45 [15.075 to 38.6125] | 22.825 [12.7625 to 40.075]
  12 weeks | 37.575 [23.6375 to 50.2] | 34.45 [18.2 to 54.2625] | 28.7 [18.2625 to 37.45]
Statistical Analysis 1: Comparison: Anakinra (Long); Paired analysis versus baseline; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Death or Hospital Admission for Heart Failure
Description: We will monitor survival and hospitalization for heart failure throughout the 24 week follow-up
Time Frame: 24 weeks
Population: All analyses were restricted to patients with a minimum of 2 weeks follow-up.
Measure: Number; unit: participants
Arm/Group | Anakinra (Short) | Anakinra (Long) | Placebo
Number analyzed (Participants) | 16 | 18 | 18
participants | 4 | 1 | 3
Statistical Analysis 1: Comparison: Anakinra (Short) vs Anakinra (Long) vs Placebo; Test type: Superiority — Log-rank test; p = 0.12, Log Rank

ADVERSE EVENTS:
Description: All analyses were restricted to patients with a minimum of 2 weeks follow-up.
Arm/Group | Anakinra (Short) | Anakinra (Long) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/18 | 1/18
Serious Adverse Events (participants affected / at risk) | 7/16 | 3/18 | 7/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (Short) (N=16) | Anakinra (Long) (N=18) | Placebo (N=18)
Death (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Stroke (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Serious infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No